CLINICAL TRIAL: NCT03314428
Title: The Effects of Gait Retraining in Runners with Knee Osteoarthritis
Brief Title: Gait Retraining for Runners with Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Hunt, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-01228
Record Dates: First submitted 2017-10-13; First posted 2017-10-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single Group cohort study
Masking Description: Data will be analyzed by an assessor blinded to date of data collection for each testing session. Following data collection, a researcher not involved with data collection or analysis will re-code data timepoints to ensure that the assessor is unaware of the timepoint each datapoint was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gait retraining (Experimental): Runners will be taught how to modify their running gait through multiple laboratory sessions and in-field training.
  Interventions: Behavioral: Gait retraining

INTERVENTIONS:
Behavioral: Gait retraining — Over a 4-week period, runners will be asked to increase their step rate to reduce knee loading during running. Specifically, they will have to increase their preferred step rate by 10% during weekly laboratory running sessions as well as during habitual running training. In the laboratory, runners will be provided with live visual/auditory biofeedback on step rate and asked to target a specific value representing 110% or preferred step rate. During their individual running sessions, runners will be wearing a GPS-enabled watch that will provide feedback on live step rate, and they will be asked to maintain the same value as in the laboratory.

SUMMARY:
Tibiofemoral osteoarthritis (TFOA) is highly prevalent in older adults, and often causes symptoms and functional limitations. Physical activity is widely advocated in people with TFOA, and running is an easy and accessible activity that provides many benefits on general health. However, running induces high knee loads, which could potentially contribute to symptoms of runners with TFOA. Previous studies have suggested that running gait modifications can help in decreasing symptoms and knee loading in runners with knee conditions. Yet, no study has been conducted in runners with TFOA. This intervention study will investigate the effects of a 4-week running gait retraining program on symptoms and running biomechanics in runners with TFOA. We hypothesize that running modifications will decrease symptoms, improve function and reduce knee loading.

ELIGIBILITY:
Inclusion Criteria:

* TFOA of Grade 2 (mild) or 3 (moderate) on the Kellgren and Lawrence scale
* report knee pain greater than or equal to 3/10 on a numerical pain rating scale (0-10) during most days of the previous month
* run at least 10 km per week for a minimum of 6 months
* declare being comfortable running on a treadmill for at least 30 minutes

Exclusion Criteria:

* history of traumatic knee injury
* neurological or inflammatory arthritic condition
* cardiovascular or cardiopulmonary disease preventing from safely performing moderate intensity running
* presence of any lower limb condition affecting running (other than TFOA)
* use of any oral or injected corticosteroids or viscosupplementation in the previous six months
* regular use of non-steroidal anti-inflammatory drugs, analgesics or knee unloading bracing devices before, during or after running
* non-English speaking

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score (KOOS) change | Baseline, 2 weeks, 4 weeks, 2 months, 3 months, 4 months
  Validated questionnaire on symptoms and functional limitations related to knee osteoarthritis. The score is expressed in percentage (0-100), with 0 representing extreme knee problems and 100 representing no knee problems.
Peak knee adduction moment impulse change | Baseline, 4 weeks, 4 months
  Validated surrogate measure of knee joint loading during movement. Expressed as Nm/kg*sec

SECONDARY OUTCOMES:
Numerical pain rating scale for pain during running change | Baseline, 2 weeks, 4 weeks, 2 months, 3 months, 4 months
  Validated scale ranging from 0 (no pain) to 10 (worst imaginable pain), in which participants rate their worst level of pain during running over the previous week.
Step rate change | Baseline, 4 weeks, 4 months
  Number of steps taken during one minute of running.
Peak knee flexion moment impulse change | Baseline, 4 weeks, 4 months
  Validated surrogate measure of knee joint loading during running. Expressed as Nm/kg*sec

OTHER OUTCOMES:
Compliance with gait retraining change | During Week 1, 2, 3 and 4 of the retraining program
  Compliance with instructions on step rate will be measured through data collected with the provided watch and a logbook. We will also monitor weekly running distance during the course of the study.
Numeric pain rating scale for usual pain change | Baseline, 2 weeks, 4 weeks, 2 months, 3 months, 4 months
  Validated scale ranging from 0 (no pain) to 10 (worst imaginable pain), in which participants rate their level of pain during their usual daily activities over the previous week.
Numeric pain rating scale for worst pain change | Baseline, 2 weeks, 4 weeks, 2 months, 3 months, 4 months
  Validated scale ranging from 0 (no pain) to 10 (worst imaginable pain), in which participants rate their worst level of pain over the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Robert H.N. Ho Research Centre, Vancouver, British Columbia, Canada